CLINICAL TRIAL: NCT00405184
Title: A Multi-centre, Open-label, Cross-over Study to Compare the Pharmacokinetics, Safety and Tolerability of Ig NextGen 10% With Intragam P in Patients With Primary Immune Deficiency (PID)
Brief Title: Ig NextGen 10% in Patients With Primary Immune Deficiency (PID)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSLCT-PID-05-22
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Primary Immune Deficiency (PID)
Keywords: PID; IVIg; IntragamP
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: IntragamP — IntragamP - dosage based on previous dose of IntragamP prior to study entry. One cycle (Cycle 0)only administered, with dosage calculation based on body weight on Day 1 of the study and must be between 0.2-0.8 g/kg body weight. IntragamP to be administered intravenously.
Drug: Ig NextGen 10% — Ig NextGen 10% - dosage based on previous dose of IntragamP in Cycle 0. Dosage calculation to use body weight on Day 1 of Cycle 1 of the study and must be between 0.2-0.8 g/kg body weight. 7 cycles administered, and patients to be dosed at 3 to 4 week intervals (in accordance with previous dosage schedule with IntragamP). Ig NextGen 10% to be administered intravenously.

SUMMARY:
This study aims to assess the safety, tolerability and pharmacokinetics of Ig NextGen 10% in patients with primary immune deficiency currently being treated with Intragam P. Eligible patients will switch from 3 to 4 weekly intravenous Intragam P therapy to receive seven cycles of Ig NextGen 10% treatment administered intravenously at three- to four-weekly intervals. Patients will be monitored on the study for up to 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PID
* = or >6 month use of Intragam P at three- or four-weekly intervals
* = or >6 month history of IgG trough levels of ≥ 5 g/L

Exclusion Criteria:

* Newly diagnosed PID within six months prior to Screening
* Known selective IgA deficiency or antibodies to IgA
* Immunosuppressive treatment other than topical and/ or inhaled steroids and/ or low dose oral steroids
* Protein-losing enteropathies, or kidney diseases
* History of malignancies of lymphoid cells
* Any of the following laboratory results at Screening:
* Serum Creatinine > 1.5 times the upper normal limit (UNL)
* AST or ALT concentration > 2.5 times the UNL
* Albumin < 25 g/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
IgG Trough Pharmacokinetics | one month

SECONDARY OUTCOMES:
Safety and tolerability, Pharmacokinetics | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Karl Bleasel, Dr, Principal Investigator — Melbourne Health
Locations (4):
- Australia (4):
  - Flinders Medical Centre, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Melbourne, Victoria

REFERENCES:
- [Result] Bleasel K, Heddle R, Hissaria P, Stirling R, Stone C, Maher D. Pharmacokinetics and safety of Intragam 10 NF, the next generation 10% liquid intravenous immunoglobulin, in patients with primary antibody deficiencies. Intern Med J. 2012 Mar;42(3):252-9. doi: 10.1111/j.1445-5994.2011.02712.x. PMID 22212346